CLINICAL TRIAL: NCT06016712
Title: The Effect of Labor on Intraocular Pressure Fluctuation in Healthy Eyes
Acronym: ELIPFHE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Jan Zapletal, Medical Doctor, Department of Obstetrics and Gynecology, Faculty Hospital Kralovske Vinohrady
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK-VP/55l012022; Internal hospital grant (Other Grant/Funding Number: Fakultni Nemocnice Kralovske Vinohrady)
Record Dates: First submitted 2023-08-08; First posted 2023-08-30 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Intraocular Pressure; Delivery
Keywords: Intraocular pressure; delivery; pregnancy; glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant (Experimental): SENSIMED Triggerfish lenses will be applied on this Arm and Intraocular pressure during active phase of delivery will be measured
  Interventions: Device: SENSIMED Triggerfish Eye Lenses

INTERVENTIONS:
Device: SENSIMED Triggerfish Eye Lenses — Contact lenses used for measuring intraocular pressure.

SUMMARY:
Glaucoma is a multifactorial disease, an important risk factor of which is increased intraocular pressure. Fluctuations in intraocular pressure are often associated with vaginal birth, although intraocular pressure during active pushing during stage II has never been measured.. The study will be conducted on a group of patients with healthy eyes on patients who have completely fine vision or have a small refractive error and are accustomed to wearing contact lenses. The measurement of intraocular pressure itself will be carried out using SENSIMED Triggerfish contact lenses, which measure pressure every 5 minutes for 30s. This period roughly corresponds to the duration of 1-2 contractions. Inclusion in the study will be offered to patients in the 35th to 37th week of pregnancy. Prior to measurement patients will be sent to an eye clinic for a detailed examination of both eyes, which includes measuring intraocular pressure. Subsequently, pregnancy checks will take place according to the standard scheme and in the standard scope. At the onset of uterine contractions, an ophthalmologic consultant will be called, which will measure intraocular pressure between contractions using the Tonopen device and put on SENSIMED Trigerfish contact lenses in combination with a local anesthetic. The patient will have these lenses until the end of the third stage of labor, i.e. 2 hours after the birth, when the lenses are removed. In the second stage of labor, continuous monitoring by a cardiotocograph will take place. Subsequently, the obtained data from the cardiotocograph and contact lenses will be evaluated and compared by a team of ophthalmologists and gynecologists, where the investigators will be able to assess the individual fluctuations in intraocular pressure depending on the individual contractions. The aim of the study is to demonstrate or disprove the risks to the glaucoma patient due to increased intraocular pressure during active pushing in combination with uterine contraction.

DETAILED DESCRIPTION:
Glaucoma is a multifactorial disease, an important risk factor of which is increased intraocular pressure. Fluctuations in intraocular pressure are often associated with vaginal birth, although intraocular pressure during active pushing during stage II has never been measured. The study will be conducted on a group of patients with healthy eyes on patients who have completely fine vision or have a small refractive error and are accustomed to wearing contact lenses. The measurement of intraocular pressure itself will be carried out using SENSIMED Triggerfish contact lenses, which measure pressure every 5 minutes for 30s. This period roughly corresponds to the duration of 1-2 contractions. Inclusion in the study will be offered to patients in the 35th to 37th week of pregnancy.Prior to measurement patients will be sent to an eye clinic for a detailed examination of both eyes, which includes measuring intraocular pressure. Subsequently, pregnancy checks will take place according to the standard scheme and in the standard scope. At the onset of uterine contractions, an ophthalmologic consultant will be called, which will measure intraocular pressure between contractions using the Tonopen device and put on SENSIMED Trigerfish contact lenses in combination with a local anesthetic. The patient will have these lenses until the end of the third stage of labor, i.e. 2 hours after the birth, when the lenses are removed. In the second stage of labor, continuous monitoring by a cardiotocograph will take place. Subsequently, the obtained data from the cardiotocograph and contact lenses will be evaluated and compared by a team of ophthalmologists and gynecologists, where the investigators will be able to assess the individual fluctuations in intraocular pressure depending on the individual contractions. The aim of the study is to demonstrate or disprove the risks to the glaucoma patient due to increased intraocular pressure during active pushing in combination with uterine contraction.

ELIGIBILITY:
Inclusion Criteria:

* physiological pregnancy
* primiparous women

Exclusion Criteria:

* multiparous women
* pathological pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 9 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fluctuation of Intraocular pressure | From start of regular contractions for the length of 24 hours (at least 2 hours after delivery if patient complies about the lenses)
  Investigators will use SENSIMED Triggerfish Lenses - contact lenses used for measuring intraocular pressure. Lenses are sending detailed description of intraocular pressure in regular time range. Measurements are then send to the software which compares all collected data.
Rate of Uterine contractions | Continuous CTG will be done during II phase of delivery and at least every 2 hours durins I phase of delivery
  Cardiotocography will be used for measuring regular uterine activity. Tocography will be used for evaluation of uterine activity compared to intraocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Studeny, prof, MD, Ph.D., Study Chair — Fakultni Nemocnice Kralovske Vinohrady
Locations (1):
- Faculty Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No